CLINICAL TRIAL: NCT00881088
Title: Prophylaxis of Venous Thromboembolism in Patients With a Nonsurgical Fracture of the Lower Extremity Immobilised in a Below-Knee Plaster Cast
Brief Title: Prophylaxis of Thromboembolic Complications Trial: Thromboprophylaxis Needed in Below Knee Plaster Cast Immobilization for Ankle and Foot Fractures
Acronym: PROTECT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Red Cross Hospital Beverwijk (Other)
Responsible Party: Principal Investigator, R.J. Derksen, Principal investigator, Red Cross Hospital Beverwijk
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROTECT
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2009-05

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Deep vein trombosis; Profylaxis; Below knee plaster cast; Ankle fracture
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Ankle Fractures | interventions — Nadroparin; Fondaparinux

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): Patients randomized to the no intervention group
- Nadroparin (Experimental): Subjects randomized to group receiving nadroparin 0,3 cc daily during immobilization
  Interventions: Drug: Nadroparin
- Fondaparinux (Experimental): Subjects randomized to fondaparinux 2,5 mg daily group during immobilization
  Interventions: Drug: Fondaparinux

INTERVENTIONS:
Drug: Nadroparin — nadroparin 0,3 cc once daily during immobilization period
  Other Names: Fraxiparin
  Arms: Nadroparin
Drug: Fondaparinux — Fondaparinux 2,5 mg daily during immobilization period
  Other Names: Arixtra
  Arms: Fondaparinux

SUMMARY:
Objective:

The purpose of this study is to determine the need for thromboprophylaxis in patients with a fracture of the lower extremity being treated conservatively in a below-knee plaster cast and to assess if both of the two tested prophylactic treatments are effective for this indication.

Hypothesis:

Nadroparine and Fondaparinux are both effective in preventing a thromboembolic event in patients with a nonsurgical fracture of a lower extremity immobilised in a below-knee plaster cast.

DETAILED DESCRIPTION:
Study Design:

A prospective, randomised, controlled, single blinded, multi-centre trial.

Intervention:

After meeting the inclusion criteria stated above and obtaining informed consent, patients will be randomly assigned to three groups: one receiving Nadroparine (2850 IE anti-Xa = 0,3 ml, given once daily), one receiving Fondaparinux (2,5 mg = 0,5 ml, given once daily) and one receiving no prophylaxis. These dosages are standard for the use in thromboprophylaxis. The first two groups will be instructed by a trained nurse in subcutaneous self-injection of the medicine and will be given pre-filled disposable syringes for once-daily administration for the duration of immobilisation.

In the light of current scientific knowledge a placebo effect of subcutaneous injections of saline in the control group is implausible since the outcome measure (colour duplex sonography) is an objective one.

Patients further will receive a letter explaining the symptoms suggesting the development of deep-vein thrombosis, pulmonary embolism and adverse events and will be asked to contact the emergency room when any of these would occur.

All patient-information will be coded so that it cannot be traced back to the individual patient. This coded information can be used for publication.

Outcome:

At the time of removal of the plaster cast symptoms or signs suggestive of DVT will be noted and a colour duplex ultrasonography of the treated limb will be performed in all patients by an experienced technician according to a strict diagnostic test protocol (see enclosure 1). When there is incompressibility of a vein or lack of flow the diagnosis of DVT is made. The technician will be blinded to treatment.

In case of a suspected pulmonary embolism pulmonary angiography will be performed.

The following risk-factors for DVT will be recorded: age, sex, body mass index (BMI), current smoking, use of estrogen-containing hormonal replacement therapy or oral contraception, active cancer (treatment on going or stopped for less than one year), congenital or acquired hypercoagulable state, previous deep venous thromboembolism and varicose veins.

Safety will be assessed as a secondary outcome. Adverse events such as haematomas, bleeding and allergic reactions will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years
* with a nonsurgical fracture of the lower extremity requiring immobilisation in a below-knee plaster cast for a minimum of 4 weeks.

Exclusion Criteria:

* Delay between injury and Emergency Department visit greater than three days
* Pregnancy/ lactation
* Body weight < 50 kg
* Severe hepatic impairment
* Severe renal impairment (creatinin-clearance < 30 ml/min)
* Known hypersensitivity to nadroparine or fondaparinux
* Pre-existing venous thromboembolism
* Pre-existing post-thrombotic syndrome
* Documented congenital or acquired bleeding tendency/disorder(s)
* Active, clinically significant bleeding
* Clinically significant bleeding within the past six months
* Previous or active bleeding from the digestive tract by peptic ulcer, tumours, hiatus hernia or diverticulosis
* Severe hypertension (systolic blood pressure above 180 mmHg or diastolic blood pressure above 110 mmHg)
* Bacterial endocarditis
* Haemorrhagic stroke within the previous two months
* Severe head injury within the previous three months
* Intraocular, spinal, and/or brain surgery within the previous twelve months
* Major surgery within the previous two months
* Treatment with LMWH or other anticoagulants
* Anticoagulant therapy required or likely to be required during the study period (e.g. planned surgery justifying pharmacological thromboprophylaxis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Estimated)
Dates: Start 2009-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure is deep vein trombosis as detected by venous duplex | subjects are assessed after 6 weeks

SECONDARY OUTCOMES:
Bleeding complications | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roelf S Breederveld, MD, PhD, Study Director — Red Cross Hospital Beverwijk; Yannick M Groutars, MD, Principal Investigator — Red Cross Hospital Beverwijk
Locations (5):
- Netherlands (5):
  - University Medical Center Nijmegen, Nijmegen, Gelderland
  - Medical Center Alkmaar, Alkmaar, North Holland
  - VU University Medical Center, Amsterdam, North Holland
  - Red Cross Hospital, Beverwijk, North Holland
  - Spaarne Hospital, Hoofddorp, North Holland

REFERENCES:
- [Derived] Bruntink MM, Groutars YME, Schipper IB, Breederveld RS, Tuinebreijer WE, Derksen RJ; PROTECT studygroup. Nadroparin or fondaparinux versus no thromboprophylaxis in patients immobilised in a below-knee plaster cast (PROTECT): A randomised controlled trial. Injury. 2017 Apr;48(4):936-940. doi: 10.1016/j.injury.2017.02.018. Epub 2017 Feb 22. PMID 28279428